CLINICAL TRIAL: NCT01695174
Title: A Pilot Study of Xifaxan in Patients With Primary Sclerosing Cholangitis
Brief Title: A Pilot Study of Xifaxan to Treat Patients With PSC
Acronym: PSC
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Jayant A. Talwalkar, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11-006516
Record Dates: First submitted 2012-09-25; First posted 2012-09-27 (Estimated); Last update posted 2014-10-15 (Estimated); Status verified 2014-10

CONDITIONS: Primary Sclerosing Cholangitis (PSC)
Keywords: Primary Sclerosing Cholangitis; Xifaxan
MeSH Terms: conditions — Cholangitis, Sclerosing | interventions — Rifaximin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Xifaxan (Experimental): Xifaxan 550 mg two times per day for three months
  Interventions: Drug: Xifaxan

INTERVENTIONS:
Drug: Xifaxan

SUMMARY:
In the current protocol, we propose the assessment of potential beneficial effects of the antibiotic Xifaxan on liver biochemistries, liver related symptoms and Mayo risk score in 15 adult and 5 pediatric patients with PSC. Adult patients will receive Xifaxan, 550 mg twice daily over a 12-week period. Pediatric patients with PSC whose weight is greater than or equal to 40 kg will receive Xifaxan, 550 mg twice daily.

ELIGIBILITY:
Inclusion criteria:

* Diagnosis of PSC established by all of the following criteria:

  * Alkaline phosphatase >1.5 times upper limit of normal for at least 6 months duration
  * Gamma-glutamyl transferase (GGT) >1.5 times upper limit of normal in pediatric patients
  * Cholangiography demonstrating intrahepatic and/or extrahepatic biliary obstruction, beading, or narrowing consistent with PSC
  * Liver histology in the past (if available for review) with features consistent with or diagnostic of PSC
* Both genders
* Adults: Ages 18-75 years.
* Pediatric: Weight > 40 kg
* Patient's informed consent for study participation

Exclusion criteria:

* Treatment with systematic antibiotics, Azulfidine, ursodeoxycholic acid, corticosteroids, colchicine, methotrexate, azathioprine, cyclosporine, chlorambucil, budesonide, pentoxifylline, tacrolimus, vitamin E or prednisone in the preceding three months
* Active drug or alcohol use
* Prior history of allergic reaction to the antibiotics which will be used in the study
* Any condition that, in the opinion of the investigator, would interfere with the patient's ability to complete the study safely or successfully
* Evidence of decompensated liver disease such as recurrent variceal bleeding, refractory ascites or spontaneous hepatic encephalopathy
* Anticipated need for transplantation in one year (Mayo survival model <80% one-year survival without transplant)
* Findings highly suggestive of liver disease of other etiology such as chronic alcoholic liver disease, chronic hepatitis B or C infection, hemochromatosis, Wilson's disease, 1-antitrypsin deficiency, non-alcoholic steatohepatitis, primary biliary cirrhosis or secondary sclerosing cholangitis
* Treatment with any study medications in the preceding three months
* Pregnancy or current lactation; subjects becoming pregnant during the study despite all the precautions will be withdrawn and referred to their primary physicians

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2012-08; Primary Completion 2013-12 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Improvement in alkaline phosphatase | Three months
  An improvement in elevated levels of alkaline phosphatase to less than half of the initial level at study entry
Absence of treatment failure | Three months
  Absence of treatment failure which is defined as any of the following: death, need for liver transplantation, side effects requiring discontinuation of therapy, worsening of liver biochemistries, voluntary discontinuation for any reason, marked worsening of fatigue or itching.

CONTACTS AND LOCATIONS:
Overall Officials: Jayant Talwalkar, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- [Result] Tabibian JH, Gossard A, El-Youssef M, Eaton JE, Petz J, Jorgensen R, Enders FB, Tabibian A, Lindor KD. Prospective Clinical Trial of Rifaximin Therapy for Patients With Primary Sclerosing Cholangitis. Am J Ther. 2017 Jan/Feb;24(1):e56-e63. doi: 10.1097/MJT.0000000000000102. PMID 24914504